CLINICAL TRIAL: NCT03892148
Title: Evaluation of an Optimization Protocol for Diuretics in the Decompensation of Chronic Heart Failure: Randomized Trial in Clusters With Sequential Permutation
Brief Title: Protocol of Diuretics Use in Congestive Therapy in Heart Failure
Acronym: ProDUCT-HF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University Hospital, Grenoble (Other); Hospices Civils de Lyon (Other); Hôpital de la Croix-Rousse (Other); CH Puy en Velay (Unknown); CH Moulins-Yzeure (Unknown); CH Riom (Unknown); Infirmerie Protestante de Lyon (Other); CH Issoire (Unknown); CH Annecy Genevois (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CHU-428; 2018-A02971-54 (Other: 2018-A02971-54)
Record Dates: First submitted 2019-02-22; First posted 2019-03-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure; Acute Heart Failure; Chronic Heart Failure
Keywords: Heart Failure; Diuretics; Diuretic resistance; Loop diuretics; Furosemide
MeSH Terms: conditions — Heart Failure | interventions — Furosemide; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard (Active Comparator): Use of loop diuretics and thiazide diuretics leaves to the discretion of the responsible physician
  Interventions: Drug: Furosemide; Drug: Hydrochlorothiazide
- Protocol (Experimental): use of loop diuretics and thiazide diuretics according to the CARRESS-HF protocol developed by the Heart Failure Network
  Interventions: Drug: Furosemide; Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Furosemide — Protocol for the use of diuretics
Drug: Hydrochlorothiazide — Protocol for the use of diuretics

SUMMARY:
The main objective of the study is to determine if a diuretic adaptation protocol in the decompensation of chronic heart failure is more effective but also safer than the current non-protocolized practice.

DETAILED DESCRIPTION:
Diuretics are the main treatment for congestive decompensation of chronic heart failure. For symptomatic purposes, the goal is to decrease the volume overload. In these patients, loop diuretics are used in high doses, sometimes in combination with other classes of diuretics such as thiazides to achieve synergistic, faster and more effective action, and to combat diuretic's resistance. This use, well known to cardiologists and based on a rich pharmacology, more than 40 years old, lacks robust scientific data in real life. Current studies are mainly based on patients with renal insufficiency or limited to cardio-renal syndrome. The CARRESS-H study in 2012 is one of them. The protocol for the use of diuretics from this study was included in 2017 as a benchmark in a publication of the NEJM. It therefore seems necessary to consider the exercise of this protocol in the management of the decompensation of chronic cardiac heart failure. There is, to the investigator's knowledge, no similar study to test this protocol as a "real life" exercise.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients hospitalized for chronic decompensated congestive heart failure without acute pulmonary edema and acute cardiac decompensation against a background of hypertensive crisis
* covered under a social security program
* with legal capacity to give voluntary informed consent to participate in the study

Exclusion Criteria:

* First episode of decompensated congestive heart failure
* Protocolized shock or hypotension (<90 mmHg blood pressure) managed or requiring nitrovasodilators or non-invasive ventilation
* One of the following cardiovascular pathologies: acute myocardial infarction / cardiac tamponade / aortic dissection / acute pulmonary embolism / heart transplant / ventricular assist device / acute pulmonary edema / hypertensive crisis
* More than 12h of intravenous diuretics administered prior to inclusion
* Generalized edema caused by cirrhosis or nephrotic syndrome
* Requiring pleural or peritoneal tap for therapeutic purposes
* Patient allergic or intolerant to furosemide and on long-term bumetanide use
* Patient in dialysis or end-stage chronic kidney disease (CKD-EPI-calculated GFR <15 mL/min/1.73m²) or acute kidney injury of known non-cardiac cause
* Severe hypokalemia (< 3 mmol/L) on admission
* Patient who is pregnant, breastfeeding, or of childbearing age not on effective contraception
* Adult patient safeguarded under court protection measures (guardianship, wardship, or judicial protection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 299 (Actual)
Dates: Start 2019-05-17 (Actual); Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Change in the serum creatinine level | at 96 hours of admission
  serum creatinine
change in weight | at 96 hours of admission
  The weight will be measured in kilograms

SECONDARY OUTCOMES:
Time of intravenous administration of diuretics | at 1 month
  Length of time of intravenous administration of diuretics in days
severity of acute kidney injury during hospitalisation | at 1 month
  Acute kidney injury requiring interruption of treatment
Severe Hypokaliemia | at month
  Severe hypokalaemia means hypokalaemia that requiring interruption of treatment, dialysis or transfer in intensive care.
Number of rehospitalization for heart failure or kidney failure | At 30 days after the date of randomisation
  Number of rehospitalization for heart failure or kidney failure
Mortality (all cause and heart failure) | At 30 days after the date of randomisation
  Number of death of participants
Dose of diuretics | At 30 days after the date of randomisation
  Comparison of diuretics dose of Furosemide and/or Thiazid diuretic. The dose will be measured on milligrams per day.
Description and comparison of global cost between the two groups | At 30 days after the date of randomisation
  Description and comparison of global cost between the two groups
Estimated plasma volume change | At 30 days after the date of randomisation
  Estimated plasma volume change captured via hemoglobin-to-hematocrit ratio (Hb/Ht) using the Strauss formula
change in bodyweight | at 96 hours after admission of patient
  The weight will be measured in kilograms
Blood chemistry (serum creatinine) | month 1
  serum creatinine
Blood chemistry (glomerular filtration rate) | month 1
  glomerular filtration rate (GFR) estimated using the CKD-EPI equation
Blood chemistry | month 1
  NT-proBNP or BNP (as available)
Blood chemistry (plasma volume estimated) | month 1
  plasma volume estimated via hemoglobin-to-hematocrit ratio (Hb/Ht)

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CLERFOND, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (9):
- France (9):
  - Ch Annecy, Annecy
  - Chu Clermont-Ferrand, Clermont-Ferrand
  - CHU de GRENOBLE, Grenoble
  - Ch Issoire, Issoire
  - CH PUY, Le Puy-en-Velay
  - Infirmerie Protestante de Lyon, Lyon
  - Ch Lyon Sud, Lyon
  - Ch Moulins, Moulins
  - CH RIOM, Riom